CLINICAL TRIAL: NCT06596161
Title: Effect or Iron Therapy on Fatigue Symptoms in Non-anemic Iron Deficient Women of Reproductive Age
Brief Title: Iron Therpay and Fatigue in Women of Reprodcutive Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Park Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPMC/IRB-No/1388; CPMC (Other: CPTH)
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Fatigue Syndrome, Chronic; Fatigue
Keywords: fatigue
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fatigue | interventions — Ferric Oxide, Saccharated

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Receiving Iron
  Interventions: Drug: Iron sucrose
- Control Group (Placebo Comparator): Receiving Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Iron sucrose — Receving iron
  Arms: Study Group
Drug: Placebo — Placebo
  Arms: Control Group

SUMMARY:
For the assessment of anemia and then assessment of fatigue levels in non-anemic women followed by assessment of iron levels and intervention of iron and placebo

ELIGIBILITY:
Inclusion Criteria:

reproductive age non-anemic fatigued

Exclusion Criteria:

anemiac males

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females of reproductive age
Enrollment: 194 (Actual)
Dates: Start 2023-02-25 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-03-02 (Actual)

PRIMARY OUTCOMES:
Fatigue Score improvemnt | 60 days
  improvement in fatigue levels

CONTACTS AND LOCATIONS:
Locations (1):
- Central Park Teaching Hospital, Lahore, Punjab Province, Pakistan